CLINICAL TRIAL: NCT01393470
Title: A Long-term Follow-up Registry-based Cohort Study of HPV Vaccine Efficacy Against Cervical Pre-cancerous Lesions and Cervical Cancers in a Cohort of Females Previously Enrolled From Finland in Study HPV-008, as Compared to a Non-intervention Population -Based Reference Cohort of Females From Finland
Brief Title: Evaluation of Long-term HPV Vaccine Efficacy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tampere University (Other)
Collaborators: FinnMedi Oy (Industry); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Matti Lehtinen, Prof., Tampere University
Other Study IDs: 115006 (HPV-027)
Record Dates: First submitted 2011-07-05; First posted 2011-07-13 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Uterine Cervical Cancer
Keywords: HPV; Vaccine; long-term efficacy; registry-based study; Evaluation of long-term HPV vaccine efficacy: a population-based, registry-based cohort study in Finland.
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cytological cervical (liquid based and/or conventional) samples. Colposcopy directed cervical biopsy samples fixed in formalin.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort A (Trial Cohort, Vaccinated during HPV-008): Cohort A subjects were previously enrolled in the HPV-008 study, and have received at least 1 dose of the HPV vaccine.
  Cohort A subjects have provided written informed consent prior to enrolment to allow retrieval of biospecimens for HPV DNA testing and confirmation of diagnosis.
  Subjects who provided written informed consent prior to enrolment for the use of their personal identifier for linkage purposes to Finnish Registries.
  Interventions: Procedure: Screening for cervical cancer
- Cohort B1 + B2: Cohort B1 subjects were previously enrolled in the HPV-008 study and received at least 1 dose of HPV vaccine as cross-over vaccination at the end of the HPV-008 study.
  Cohort B1 subjects have provided written informed consent prior to enrolment to allow retrieval of biospecimens for HPV DNA testing and confirmation of diagnosis.
  Subjects who provided written informed consent prior to enrolment for the use of their personal identifier for linkage purposes to Finnish Registries.
  Cohort B2 (Trial Cohort, Non-Vaccinated)
  Interventions: Procedure: Screening for cervical cancer
- Cohort C (Referent Cohort, Non-Vaccinated): Cohort C subjects have not participated in the HPV-008 study but have been enrolled in the Referent Cohort.
  Cohort C subjects have not received any HPV vaccination (neither Cervarix, nor Gardasil, nor any experimental HPV vaccine).
  Cohort C subjects are partially matched to HPV-008 in terms of the geographical recruitment area.
  Subjects who provided written informed consent prior to enrolment for the use of their personal identifier for linkage purposes to Finnish Registries.
  Interventions: Procedure: Screening for cervical cancer

INTERVENTIONS:
Procedure: Screening for cervical cancer — Organized screening for cervical cancer start for all cohorts at the age of 25 years with 5 year interval.

SUMMARY:
Summary

For ethical and practical reasons pre-licensure clinical efficacy phase III trials for GSK Biologicals' HPV-16/18 LI VLP AS04 vaccine used cervical intraepithelial grade 2 and above (CIN2+) lesions as surrogate efficacy endpoint for cervical cancer. The long-term impact of HPV vaccination on cervical cancer as well as other HPV-related non- cervical cancers is, however, an area warranting further exploration in the post-licensure setting. Results of the multinational phase III trial demonstrated high vaccine efficacy against CIN2+ associated with HPV-16 and/or HPV-18, significant vaccine efficacy against CIN2+ and CIN3+ irrespective of HPV type in the lesion as well as evidence of protection against CIN2+ associated with HPV types 31 and 45 [Paavonen, et al. 2009]. Over time, vaccinated cohorts should benefit from a substantial reduction in the incidence of cervical cancer considering impact on oncogenic non-vaccine HPV types. This long-term study is conducted to evaluate the long-term impact of GSK Biologicals' HPV-16/18 vaccine on the occurrence of cervical pre-cancerous lesions and cervical cancer with the following objectives:

* To assess the long-term efficacy of the HPV-16/18 L1 VLP AS04 vaccine on the occurrence of cervical cancer including its immediate precursors (CIN3+): cervical intraepithelial neoplasia grade 3 (CIN3) and adenocarcinoma in situ (AIS) by comparing cohorts A and C (see below).
* To assess the efficacy of HPV-16/18 L1 VLP AS04 vaccine on the occurrence of the following potentially HPV related non-cervical cancers such as vulvar intraepithelial neoplasia, vaginal intraepithelial neoplasia, anogenital neoplasia and oropharyngeal neoplasia by comparing cohorts A and C (see below)
* To assess as an explanatory objective the occurrence of CIN3+ breakthrough cases associated with HPV-16 or HPV-18 infection in subjects vaccinated with HPV-16/18 L1 VLP AS04 vaccine by close surveillance of cohorts and cross vaccinated cohort B (see below)

This prospective, observational cohort study is undertaken in originally 16-17 year-old Finnish females who have participated in the GSK Biologicals' HPV-008 trial (NCT00122681) with regular clinical follow-up, and can be divided in Cohort A: Female subjects from Finland who received HPV-16/18 L1 VLP AS04 vaccine in the HPV-008 study between May 2004 and May 2005 (N=2409), and Cohort B: Female subjects from Finland who received the Hepatitis A control vaccine in the HPV-008 study (N=2399). All subjects were offered the HPV-16/18 L1 VLP AS04 vaccine or screening for cervical cancer at the end of the study (age 21-22): 50% of the subjects, chose not to take cross-over HPV vaccination at HPV-008 study end. Referent Cohort C: A population-based reference cohort of female subjects from Finland who have not been exposed to any HPV vaccine (either during a HPV vaccine trial, or commercially available vaccine; i.e. Cervarix or Gardasil), enrolled in this study in May - September 2003 or May - September 2005, altogether 15536 subjects).

Prospective data collection will start at the HPV screening invitation for each subject in 2013. Several analyses are planned including an analysis at 8 years post-completion of the HPV-008 study (by 2020) and will provide a total evaluation time of approximately 15 years since first vaccination in the Cohort A.

The study is self-contained for the primary and secondary endpoints. Data from the HPV-008 trial will be used to address exploratory objectives mentioned above. Data collection will be performed using the databases from the University of Tampere.

ELIGIBILITY:
Inclusion Criteria:

* Trial Cohort (16-17 years at baseline) - the cohort of Finnish subjects who participated in the GSK Biologicals' HPV-008 trial (NCT00122681):
* Cohort A: subjects who received HPV-16/18 L1 VLP AS04 vaccine between May 2004 and May 2005.
* Cohort B: subjects who received the Hepatitis A control vaccine. All subjects were offered the HPV-16/18 L1 VLP AS04 vaccine at the end of the study (age 21-22).
* Cohort B1: subjects who received the Hepatitis A control vaccine and then received cross-over HPV vaccination at HPV-008 study end.
* Cohort B2: subjects who received the Hepatitis A control vaccine and who did not receive cross-over HPV vaccination at HPV-008 study end.
* Referent cohort (18-19 years at baseline):
* Cohort C: A population-based reference cohort of female subjects from Finland who have not been exposed to any HPV vaccine enrolled in this study in May 2005, immediately after recruitment of the HPV-008 clinical trial subjects had been stopped (approximately 9,000 subjects).

Exclusion Criteria:

* Trial Cohort (Cohort A and B): Previous or planned administration of an HPV vaccine not foreseen by the HPV-008 study protocol or any HPV-008 extension study protocol (Gardasil or any experimental HPV vaccine).
* Referent cohort (Cohort C): Previous or planned administration of an HPV vaccine (Cervarix, Gardasil or any experimental HPV vaccine).

Ages: 16 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Trial Cohort (16-17 years at baseline) - the cohort of Finnish subjects who participated in the GSK Biologicals' HPV-008 trial (NCT00122681):
  Cohort A: subjects who received HPV-16/18 L1 VLP AS04 vaccine between May 2004 and May 2005.
  Cohort B: subjects who received the Hepatitis A control vaccine. All subjects were offered the HPV-16/18 L1 VLP AS04 vaccine at the end of the study (age 21-22):
  Cohort B1: subjects who received the Hepatitis A control vaccine and then received cross-over HPV vaccination at HPV-008 study end.
  Cohort B2: subjects who received the Hepatitis A control vaccine and who did not receive cross-over HPV vaccination at HPV-008 study end.
  Referent cohort (18-19 years at baseline):
  Cohort C: A population-based reference cohort of female subjects from Finland who have not been exposed to any HPV vaccine enrolled in this study in May 2005, immediately after recruitment of the HPV-008 clinical trial subjects had been stopped (approximately 9,000 subjects).
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2011-05; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of intraepithelial neoplasia grade 3 or worse (CIN3+). including CIN3, cervical cancer (squamous cell carcinoma or adenocarcinoma). | The time frame is up to 15 years (for the interim analyses: 4, 7 and 10 years). (Start and end of passive follow-up, Cohorts A and B: 01.01.2010 - 31.12. 2024; Cohorts C1 and C2: 01.10.2007/01.10.2008 - 30.09.2021/30.09.2023.)
  To estimate the long-term vaccine efficacy by comparing the incidence rate of cervical cancers and pre-cancerous lesions (CIN3+) in Cohort A vs. Cohort C.

SECONDARY OUTCOMES:
Occurrence of potentially HPV related non-cervical cancers or pre cancerous lesions, including but not limited to the occurrence of vulvar intraepithelial neoplasia and vaginal intraepithelial neoplasia. | The time frame for the objectives of the study is up to 15 years. (Start and end of passive follow-up, Cohorts A and B: 01.01.2010 - 31.12. 2024; Cohorts C1 and C2: 01.10.2007/01.10.2008 - 30.09.2021/30.09.2023.)
  To estimate the efficacy of HPV-16/18 vaccine against non-cervical cancers by comparing the incidence of non-cervical cancers in Cohort A vs. Cohort C.

CONTACTS AND LOCATIONS:
Overall Officials: Matti Lehtinen, M.D., Ph.D., Principal Investigator — Tampere University
Locations (15):
- Finland (15):
  - Väestöliitto Seksuaaliterveysklinikka, Helsinki
  - Nuorten rokotetutkimukset, Jyväskylä
  - Nuorten rokotetutkimukset, Kotka
  - Nuorten rokotetutkimukset, Kouvola
  - Nuorten rokotetutkimukset, Kuopio
  - Nuorten rokotetutkimukset, Lahti
  - Nuorten rokotetutkimukset, Lappeenranta
  - Nuorten rokotetutkimukset, Mikkeli
  - VL-Medi Oy/Pikkuklinikka, Oulu
  - Nuorten rokotetutkimukset, Pori
  - Nuorten rokotetutkimukset, Rauma
  - Nuorten rokotetutkimukset, Seinäjoki
  - Nuorten rokotetutkimukset, Tampere
  - Nuorten rokotetutkimukset, Turku
  - Nuorten rokotetutkimukset, Vaasa

REFERENCES:
- [Background] Paavonen J, Naud P, Salmeron J, Wheeler CM, Chow SN, Apter D, Kitchener H, Castellsague X, Teixeira JC, Skinner SR, Hedrick J, Jaisamrarn U, Limson G, Garland S, Szarewski A, Romanowski B, Aoki FY, Schwarz TF, Poppe WA, Bosch FX, Jenkins D, Hardt K, Zahaf T, Descamps D, Struyf F, Lehtinen M, Dubin G; HPV PATRICIA Study Group. Efficacy of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine against cervical infection and precancer caused by oncogenic HPV types (PATRICIA): final analysis of a double-blind, randomised study in young women. Lancet. 2009 Jul 25;374(9686):301-14. doi: 10.1016/S0140-6736(09)61248-4. Epub 2009 Jul 6. PMID 19586656
- [Background] Paavonen J, Jenkins D, Bosch FX, Naud P, Salmeron J, Wheeler CM, Chow SN, Apter DL, Kitchener HC, Castellsague X, de Carvalho NS, Skinner SR, Harper DM, Hedrick JA, Jaisamrarn U, Limson GA, Dionne M, Quint W, Spiessens B, Peeters P, Struyf F, Wieting SL, Lehtinen MO, Dubin G; HPV PATRICIA study group. Efficacy of a prophylactic adjuvanted bivalent L1 virus-like-particle vaccine against infection with human papillomavirus types 16 and 18 in young women: an interim analysis of a phase III double-blind, randomised controlled trial. Lancet. 2007 Jun 30;369(9580):2161-2170. doi: 10.1016/S0140-6736(07)60946-5. PMID 17602732
- [Background] Lehtinen M, Idanpaan-Heikkila I, Lunnas T, Palmroth J, Barr E, Cacciatore R, Isaksson R, Kekki M, Koskela P, Kosunen E, Kuortti M, Lahti L, Liljamo T, Luostarinen T, Apter D, Pukkala E, Paavonen J. Population-based enrolment of adolescents in a long-term follow-up trial of human papillomavirus vaccine efficacy. Int J STD AIDS. 2006 Apr;17(4):237-46. doi: 10.1258/095646206776253453. PMID 16595046
- [Background] Lehtinen M, Paavonen J. Effectiveness of preventive human papillomavirus vaccination. Int J STD AIDS. 2003 Dec;14(12):787-92. doi: 10.1258/095646203322556084. PMID 14678583
- [Background] Lehtinen M, Apter D, Dubin G, Kosunen E, Isaksson R, Korpivaara EL, Kyha-Osterlund L, Lunnas T, Luostarinen T, Niemi L, Palmroth J, Petaja T, Rekonen S, Salmivesi S, Siitari-Mattila M, Svartsjo S, Tuomivaara L, Vilkki M, Pukkala E, Paavonen J. Enrolment of 22,000 adolescent women to cancer registry follow-up for long-term human papillomavirus vaccine efficacy: guarding against guessing. Int J STD AIDS. 2006 Aug;17(8):517-21. doi: 10.1258/095646206778145550. PMID 16925896